CLINICAL TRIAL: NCT04058574
Title: Measurement and Relationships of Proprioceptive Isokinetic Repositioning With Muscle Strength, Functional Testing, and Self-reported Questionaires Before and After Anterior Cruciate Ligament Reconstruction: A Prospective Study With 12-months Post Operative Follow-up.
Brief Title: Proprioceptive Isokinetic Repositioning, Functional Testing, and a Self-reported Questionnaire Before and After Anterior Cruciate Ligament Reconstruction
Acronym: PRO-ACL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Caen (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Principal Investigator, Joffrey DRIGNY, Chief Resident PM&R and Sport departments MD, MSc, University Hospital, Caen
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PRO-ACL
Record Dates: First submitted 2019-08-09; First posted 2019-08-15 (Actual); Last update posted 2020-07-15 (Actual); Status verified 2020-07

CONDITIONS: ACL Tear; ACL - Anterior Cruciate Ligament Deficiency
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Intervention Model Description: Intervention Group "ACL": 30 patient, athletes, with ACL deficiency candidate to a surgical ACL reconstruction Control Group: 15 healthy volunteers, athletes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ACL (Active Comparator): Intervention Group "ACL": 30 patient, athletes, with ACL deficiency candidate to a surgical ACL reconstruction
  Interventions: Device: Proprioception measurement on isokinetic dynamometer
- Control (Placebo Comparator): Control Group: 15 healthy volunteers, athletes.
  Interventions: Device: Proprioception measurement on isokinetic dynamometer

INTERVENTIONS:
Device: Proprioception measurement on isokinetic dynamometer — Proprioception measurement on isokinetic dynamometer using joint position sense (JPS) and the threshold to detection of passive motion (TTDPM)

SUMMARY:
This prospectively study aims to evaluate the evolution of knee joint proprioception on isokinetic dynamometer before and after Anterior Cruciate Ligament (ACL) reconstruction and its relationships with muscle strength, self reported questionnaire and return to sport. This study will include 30 athletes with isolated ACL rupture, and treated with ACL reconstruction surgery and 15 healthy volunteers.

DETAILED DESCRIPTION:
Anterior cruciate ligament (ACL) rupture is a common injury in athletes. It has multiple consequences on the knee: instability, pain, loss of muscle strength, proprioceptive impairments, modification of the knee kinematics and premature knee osteoarthritis. In athletes, the majority of these injuries are treated with ACL reconstruction surgery. The main objective of this treatment is the reduction of knee instability to allow return to sport, and this at the same level prior to the injury. Thus, the athlete's follow-up after the surgery is essential to guide the return to sport and to ensure that the knee sensorimotor control allows the return to sport. Currently this assessment is based primarily on functional testings and measurement of muscle strength.

The investigators propose to prospectively study the evolution of instrumentally measured knee proprioception using isokinetic dynamometer before and after ACL reconstruction as well as a study of the factors associated with its favorable evolution and its impact in the return to sport and its level.

ELIGIBILITY:
Inclusion Criteria:

* Isolated and primary tear of the ACL
* Individual candidate for an ACL reconstruction surgery.
* Acute ACL injury (<6 weeks)
* Athletes (person who competes in one or more sports that involve physical strength, speed or endurance) whatever their level of sport practice
* Internet access

Exclusion Criteria:

* Prior knee surgery
* Complex ligamentous lesion (lateral ligaments, posterior cruciate ligament)
* Surgery for meniscal lesions (patients initially included but warranting meniscal surgery during arthroscopy will be secondarily excluded from the study.)
* Recent muscle damage
* History of significant injury on the healthy knee
* ACL rupture recurrence
* Pregnant woman
* Neurological or vestibular antecedent with sequelae
* Individuals taking treatment altering alertness (neuroleptics, sedatives)
* Informed consent not obtained

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2021-09-01 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline passive proprioceptive evaluation after 7 months | ACL group: 6 weeks after surgery and 7 months after surgery; Healthy group: one evaluation at a single point in time through study completion, an average of 1 year
  Measurement of knee proprioception by the passive repositioning technique (JPS, in degrees) on isokinetic dynamometer.
Change from Baseline active proprioceptive evaluation after 7 months | ACL group: 6 weeks after surgery and 7 months after surgery; Healthy group: one evaluation at a single point in time through study completion, an average of 1 year
  Measurement of knee proprioception by the active repositioning technique (JPS, in degrees) on isokinetic dynamometer.
Change from Baseline TDPM (Threshold to Detection of Passive Motion) evaluation after 7 months | ACL group: 6 weeks after surgery and 7 months after surgery; Healthy group: one evaluation at a single point in time through study completion, an average of 1 year
  Measurement of knee proprioception by the Threshold to Detection of Passive Motion (TDPM in degrees) on isokinetic dynamometer.

SECONDARY OUTCOMES:
Strength | ACL group: Two evaluations on both injured and healthy knees: (1) 3 months after surgery and (2) 7 months after surgery; Healthy group: one evaluation at a single point in time through study completion, an average of 1 year
  Measurement of knee extensors and flexors peak strength (in newton.meter, Nm) on isokinetic dynamometer.
ACL-RSI questionnaire (Anterior Cruciate Ligament-Return to Sport after Injury) | ACL group: Four evaluations on both injured and healthy knees: (1) 2 weeks before surgery, (2) 3 months after surgery, (3) 7 months after surgery and (4) 12 months after surgery
  The ACL-RSI measures the patient's understanding of his knee. It comprises 12 questions with a score of 1 to 10 for each
Functional testing | ACL group: Two evaluations on both injured and healthy knees: (1) 3 months after surgery and (2) 7 months after surgery; Healthy group: one evaluation at a single point in time through study completion, an average of 1 year
  Hop test. Single hop: Patients are instructed to stand on one leg and perform 1 jump as far as possible, landing on the same leg.
  The total distance is recorded (in cm) .Triple hop: Patients are instructed to stand on one leg and perform 3 hops as far as possible, landing on the same leg.
  The total distance for 3 consecutive hops is recorded (in cm). Cross-over hop test : The patient hops forward 3 times while alternately crossing over a marking The patient is instructed to position themselves such that the first of the 3 hops was lateral with respect to the direction of crossover The total distance hopped forward is recorded (in cm)

CONTACTS AND LOCATIONS:
Locations (1):
- Caen University Hospital, Caen, France

IPD SHARING:
Plan to Share IPD: Undecided